CLINICAL TRIAL: NCT01337232
Title: Building Complex Language: Effect of Treatment and Dosage
Brief Title: Building Complex Language
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Governors State University (Other)
Collaborators: Rush University (Other)
Responsible Party: Principal Investigator, Catherine Balthazar, Chair, Department of Communication Disorders, Governors State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R15DC011165-01 (NIH)
Record Dates: First submitted 2011-04-13; First posted 2011-04-18 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Language Development Disorders; Learning Disorders
Keywords: language development disorders; learning disorders; sentences; syntax; school-age; language
MeSH Terms: conditions — Language Development Disorders; Learning Disabilities; Language

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 session per week (Active Comparator)
  Interventions: Behavioral: Complex sentence treatment protocol
- 2 sessions per week (Experimental)
  Interventions: Behavioral: Complex sentence treatment protocol

INTERVENTIONS:
Behavioral: Complex sentence treatment protocol — Treatment: listening, speaking, reading, and writing activities that teach three types of complex sentences. Individual sessions are 40 minutes in length, delivered by or under the supervision of a certified, trained speech-language pathologist.

SUMMARY:
This study is designed to examine how much therapy is needed in order to make significant gains in knowledge and use of complex sentences. Students will be randomly placed in individual treatment sessions that take place either once or twice per week for nine weeks. All will receive the same type of treatment, which consists of a focused series of oral and written language activities. While it is anticipated that students in both groups will benefit from treatment, we hypothesize that the twice-weekly session frequency will have a significantly greater impact on level of performance and maintenance of skills after treatment.

DETAILED DESCRIPTION:
The objective of this project is to examine outcomes of a treatment intervention designed to increase functional use of complex (multi-clausal) sentences in school-age students with primary language impairments that impact literacy and academic achievement. The treatment protocol includes: (1) three types of complex sentences (adverbial, relative, object complement), (2) encounters with complex sentences in real texts and across all modalities (speaking, listening, reading, writing, and (3) activities that engage metalinguistic understanding of complex sentences. Specific objectives are to (1) document treatment effect in terms of size and scope of impact in decontextualized as well as naturalistic language contexts, (2) document the effect of treatment intensity (dosage), (3) explore effects of sentence complexity subtype and treatment outcomes, and (4) explore relationships between treatment outcomes and participant variables (pre-treatment knowledge of complex sentences, verbal working memory, and non-verbal cognition).

The study will utilize two designs. Approximately 10 participants per year will complete the treatment, randomly assigned to one of two treatment levels. As each participant finishes, efficacy and effect size will be measured using a multiple-baseline single-subject design. Once all 30 participants have completed the treatment, effect size and the impact of dosage (treatment intensity) will be evaluated using a pretest-posttest group design, and correlations between participant characteristics and individual patterns of performance will be carefully described and analyzed.

This study targets school-age students with a Speech-Language Impairment and/or a Specific Learning Disability between the ages of 10 and 14 who are receiving services from a Speech-Language Pathologist (SLP) for one or more higher-level language behaviors. It is expected that participants will demonstrate higher levels of fluency with complex sentences compared with pretreatment baseline levels and that treatment effects will be reflected in several modalities and in naturalistic language contexts.

ELIGIBILITY:
Inclusion Criteria:

* Disability: documented language or learning disorder
* Nonverbal IQ within 1 standard deviation of mean for age
* Oral language score 1 or more standard deviations below mean for age
* Problem areas: difficulty with language in any of the following areas - reading comprehension, writing, following verbal instructions, verbal expression

Exclusion Criteria:

* hearing impairment
* autism spectrum disorder
* developmental delay
* genetic syndrome
* brain injury
* cerebral palsy
* seizure disorder

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2011-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Changes in Scores on Norm-Referenced and Criterion-Referenced Language Tests | within one month post treatment
  A battery of language comprehension and production measures given pre-treatment will be administered again following treatment. The measures include broad norm-referenced oral and written language tests and a specific criterion-referenced measure of complex sentence production.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine H Balthazar, PhD, Principal Investigator — Governors State University; Cheryl M Scott, PhD, Principal Investigator — Rush University Medical Center
Locations (2):
- United States (2):
  - Rush University Medical Center, Chicago, Illinois
  - Governors State University, University Park, Illinois